CLINICAL TRIAL: NCT00618410
Title: Intranasal CO2 for Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Capnia, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Naclerio, MD, University of Chicago
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 15835A
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2013-12

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbon dioxide (Active Comparator): nasal Carbon dioxide, USP (CO2) administered 30 minutes prior to nasal challenge
  Interventions: Device: Carbon dioxide, USP
- Placebo (Placebo Comparator): nasal placebo administered 30 minutes prior to nasal challenge
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Carbon dioxide, USP — Carbon dioxide (CO2) delivered via a nosepiece at a flow rate of 0.5 (± 0.05) SLPM for 10 seconds /nostril
  Arms: Carbon dioxide
Other: Placebo — Nasal placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to better understand the way in which CO2 (carbon dioxide) affects the symptoms of allergic rhinitis or hayfever.

Our intent is to determine if CO2 has an effect on nasal challenge with antigen as a predictor of whether it will have a beneficial effect on the treatment of seasonal allergic rhinitis.

DETAILED DESCRIPTION:
Study design: We performed a randomized, two-way crossover study in subjects with seasonal allergic rhinitis out of season. Subjects came to the Nasal Physiology Laboratory for screening, where they completed an allergy questionnaire and underwent skin-prick testing for confirmation of a grass or ragweed allergy. The skin test included positive and negative controls and the results were graded compared with the controls as 1+ to 4+ (1+: wheal larger than negative control and smaller than positive control; 2+: wheal 5-7 mm; 3+: wheal 7-10 mm; 4+: any reaction with a wheal >10 mm or pronounced pseudopodia). Subjects with positive skin test (between 2+ and 4+) and a positive history of allergic symptoms during the relevant seasons then underwent a screening nasal challenge with either grass or ragweed allergen. Subjects who passed the screening challenge (twofold increase in either ipsilateral or contralateral nasal secretions after allergen challenge compared with diluent) had a 2-week washout period and returned to the laboratory, where they were randomized to receive intranasal treatment with either CO2 or no treatment. Thirty minutes after treatment, subjects underwent a nasal challenge with allergen. Seven subjects were challenged with ragweed and five subjects were challenged with grass. Subjects had another 2-weeks washout period and were then crossed over to the other treatment followed by a similar challenge. Previous work in our laboratory using a similar challenge system showed that allergen-induced inflammatory changes are back to baseline 2 weeks after the challenge.

Subjects: Twelve subjects participated. Subjects were studied outside their allergy season. All subjects were healthy except for mild asthma requiring only as-needed bronchodilators. They were not on any medications and had not received antihistamines or leukotriene receptor antagonists for at least 1 week and intranasal steroids for at least 1 month before enrollment and for the duration of the study.

Treatment: CO2 was applied for 10 seconds in each nostril using a special applicator (plastic tight-seal nosepiece) attached to a CO2 canister and a flow control valve. It was delivered at a flow rate of 0.5 standard L/min with the mouth open to prevent inhalation. Thus, for 20-second duration of administration, the total dose of CO2 delivered was 167 mL. The amount of CO2 delivered to the mucosa is unknown. The no-treatment arm involved placement of the device but no gas was delivered. Therefore, neither the subjects nor the investigators were blinded to the treatment administered. The no-treatment arm did not involve the delivery of air without CO2 to the nose because we were concerned that blowing dry air into the nose might cause a mucosal reaction that could confound the results. We have previously shown that cold, dry air challenges create a hyperosmolar environment, triggers mast cell activation, and induces a nasonasal reaction.7 Thus, because our primary outcome was the objective measure of the nasonasal reflex, we avoided this possibility.

Nasal Challenge: The subjects were allowed 15 minutes to acclimatize to the laboratory environment before challenge. Baseline sneezes reflecting the 15 minutes of acclimatization and nasal and eye symptoms were recorded followed by collection of a nasal scraping for quantitation of eosinophils in nasal secretions. Sneezes were recorded by the subjects during each of the assessed intervals of the challenge protocol. The subjects were reminded to keep track of the number of sneezes by the research coordinator who was present for the duration of the challenges. Intranasal CO2 or sham was then applied for 10 seconds to each nostril. Thirty minutes later, sneezes and symptoms were recorded again, to reflect the 30-minute time period, and nasal challenge was initiated. Because we were interested in evaluating the effect of the treatment on allergen-induced nasal reflexes, we used filter paper disks to perform the challenges and monitor the secretory response as previously described.

Briefly, 8-mm filter paper disks (Shandon, Inc., Pittsburgh, PA) were used for both nasal challenge and collection of resultant secretions. They were placed on the anterior nasal septum, beyond the mucocutaneous junction, under direct vision using a nasal speculum, forceps, and a headlight. Fifty microliters of challenge solutions were placed on the disks, which were then applied to the nasal septum for 1 minute. Thirty seconds after removal, two preweighed filter paper disks were placed on both sides of the nasal septum for 30 seconds, collecting nasal secretions from the challenge site (ipsilateral) and the contralateral nostril. These disks were then immediately placed back into microtubes and weighed. The difference in their weight before and after challenge was the weight of produced nasal secretions, which was recorded in milligrams. Ten minutes after each challenge, the number of sneezes as well as symptoms on each side were recorded by the subjects reflective of the 10-minute interval The first challenge was performed using phenol-buffered saline, the diluent for the allergen extracts, and this was followed by 2 increasing doses of grass or ragweed allergen. The time from treatment administration to the first allergen challenge was approximately 40 minutes and to the second allergen challenge, 50 minutes. The amount of allergen applied on the paper disks for challenge were 333 and 1000 BAU (bioequivalent allergy unit) of grass allergen extract (Hollister-Stier, Spokane, WA) or 50 microliters of ragweed antigen extract at concentrations of 1:666 and 1:200 w/v (Hollister-Stier). The subjects came back to the laboratory 24 hours later and underwent a scraping of their nasal secretions to evaluate for eosinophil influx.

ELIGIBILITY:
Inclusion Criteria

1. Males and females between 18 and 45 years of age.
2. History of grass and/or ragweed allergic rhinitis.
3. Positive skin test to grass and/or ragweed antigen.
4. Positive response to screening nasal challenge.

Exclusion Criteria

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Upper respiratory infection within 14 days of study start.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Naclerio, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Baroody FM, Gavanescu L, Wang JH, DeTineo M, Naclerio RM. The effect of intranasal carbon dioxide on the acute response to nasal challenge with allergen. Allergy Asthma Proc. 2011 May-Jun;32(3):206-12. doi: 10.2500/aap.2011.32.3442. PMID 21703101

RESULTS

PARTICIPANT FLOW:
Groups:
- Carbon Dioxide, Then Placebo: Intervention sequence:
  1. Intervention #1: nasal Carbon dioxide, USP (CO2) administered 30 minutes prior to nasal challenge
  2. Intervention #2: nasal placebo administered 30 minutes prior to nasal challenge
- Placebo, Then Carbon Dioxide: Intervention sequence:
  1. Intervention #1: nasal placebo administered 30 minutes prior to nasal challenge
  2. Intervention #2: nasal Carbon dioxide, USP (CO2) administered 30 minutes prior to nasal challenge
Period: First Intervention
Arm/Group | Carbon Dioxide, Then Placebo | Placebo, Then Carbon Dioxide
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Washout Period (2 Weeks)
Arm/Group | Carbon Dioxide, Then Placebo | Placebo, Then Carbon Dioxide
Started | 7 | 6
Completed | 7 | 5
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Second Intervention
Arm/Group | Carbon Dioxide, Then Placebo | Placebo, Then Carbon Dioxide
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Study population includes subjects receiving interventions in either order.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.69 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Diluent Challenge Contralateral Secretion Weight at Antigen Challenge
Description: Fifty microliters of challenge solutions were placed on the disks, which were then applied to the nasal septum for 1 minute. Thirty seconds after removal, two preweighed filter paper disks were placed on both sides of the nasal septum for 30 seconds, collecting nasal secretions from the challenge site (ipsilateral) and the contralateral nostril. These disks were then immediately placed back into microtubes and weighed. The difference in their weight before and after challenge was the weight of produced nasal secretions, which was recorded in milligrams. Contralateral secretion weight for the diluent challenge was subtracted from that of the antigen challenge to compute this primary outcome measure.
Time Frame: 10 minutes post diluent challenge and 10 minutes post antigen challenge
Population: Excludes one patient who did not complete the second crossover intervention.
Measure: Median (Full Range); unit: milligrams
Arm/Group | Carbon Dioxide | Placebo
Number analyzed (Participants) | 12 | 12
milligrams | 6 [-3.1 to 54.1] | 19.6 [0 to 55.2]

2. Secondary Outcome: Change From Diluent Challenge Ipsilateral Secretion Weight at Antigen Challenge
Description: Fifty microliters of challenge solutions were placed on the disks, which were then applied to the nasal septum for 1 minute. Thirty seconds after removal, two preweighed filter paper disks were placed on both sides of the nasal septum for 30 seconds, collecting nasal secretions from the challenge site (ipsilateral) and the contralateral nostril. These disks were then immediately placed back into microtubes and weighed. The difference in their weight before and after challenge was the weight of produced nasal secretions, which was recorded in milligrams. Ipsilateral secretion weight for the diluent challenge was subtracted from that of the antigen challenge to compute this primary outcome measure.
Time Frame: 10 minutes post diluent challenge and 10 minutes post antigen challenge
Population: Excludes one patient who did not complete the second crossover intervention.
Measure: Median (Full Range); unit: milligrams
Arm/Group | Carbon Dioxide | Placebo
Number analyzed (Participants) | 12 | 12
milligrams | 9 [-4.8 to 90.4] | 32.6 [0 to 49.7]

3. Secondary Outcome: Change From Diluent Challenge Ipsilateral Histamine Level at Antigen Challenge
Description: After collection of nasal secretions after diluent or antigen challenge, the filter paper disks were replaced in Eppendorf tubes and the disk/tube combination was weighed to record produced secretions. Three hundred microleters of 0.9% sodium chloride solution was then placed in the tubes and mediators were allowed to elute from the disks for 24 hours at 4 degrees Celsius. The eluate was then transferred to tubes and stored at -20 degrees Celsius until assayed for histamine.
  Histamine was assayed by ELISA (Oxford Biomedical Research, Oxford, MI). The lower limit of detection of the assay is 2.5 ng/mL and samples below the detection limit were arbitrarily assigned a value of 1.25 ng/mL. The ipsilateral measure was taken from the challenge site.
  The number reported in this outcome measure was calculated by subtracting the ipsalateral histamine level at diluent challenge from the analogous measure recorded after antigen challenge. Values may be positive or negative.
Time Frame: 10 minutes post diluent challenge and 10 minutes post antigen challenge
Population: Excludes one patient who did not complete the second crossover intervention.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Carbon Dioxide | Placebo
Number analyzed (Participants) | 12 | 12
ng/mL | 0 [-2.7 to 16.6] | 2.04 [0 to 10.4]

4. Secondary Outcome: Change From Diluent Challenge Contralateral Histamine Level at Antigen Challenge
Description: After collection of nasal secretions after diluent or antigen challenge, the filter paper disks were replaced in Eppendorf tubes and the disk/tube combination was weighed to record produced secretions. Three hundred microleters of 0.9% sodium chloride solution was then placed in the tubes and mediators were allowed to elute from the disks for 24 hours at 4 degrees Celsius. The eluate was then transferred to tubes and stored at -20 degrees Celsius until assayed for histamine.
  Histamine was assayed by ELISA (Oxford Biomedical Research, Oxford, MI). The lower limit of detection of the assay is 2.5 ng/mL and samples below the detection limit were arbitrarily assigned a value of 1.25 ng/mL. The ipsilateral measure was taken from the challenge site.
  The number reported in this outcome measure was calculated by subtracting the contralateral histamine level at diluent challenge from the analogous measure recorded after antigen challenge. Values may be positive or negative.
Time Frame: 10 minutes post diluent challenge and 10 minutes post antigen challenge
Population: Excludes one patient who did not complete the second crossover intervention.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Carbon Dioxide | Placebo
Number analyzed (Participants) | 12 | 12
ng/mL | 0 [-1.2 to 1.7] | 0 [0 to 9.1]

5. Secondary Outcome: Eosinophil Influx [Pre-allergen]
Description: The number of eosinophils per 200 white blood cells was counted for each nasal secretion scraping. The percentage of eosinophils was recorded.
Time Frame: before antigen challenge
Measure: Median (Full Range); unit: percentage of white blood cells
Arm/Group | Carbon Dioxide | Placebo
Number analyzed (Participants) | 12 | 12
percentage of white blood cells | 0 [0 to 0] | 0 [0 to 2]

6. Secondary Outcome: Eosinophil Influx [Post-allergen]
Description: as for outcome 5
Time Frame: after antigen challenge
Measure: Median (Full Range); unit: percentage of white blood cells
Arm/Group | Carbon Dioxide | Placebo
Number analyzed (Participants) | 12 | 12
percentage of white blood cells | 0 [0 to 31] | 0 [0 to 4]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Carbon Dioxide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes